CLINICAL TRIAL: NCT06018181
Title: Outcomes After Intravenous Alteplase / Tenecteplase With or Without Shuxuetong Injection in Routine Clinical Practice: A Patient Registry
Brief Title: Outcomes After Intravenous Alteplase / Tenecteplase With or Without Shuxuetong Injection in Routine Clinical Practice
Status: Recruiting | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, MD, PhD, Dongzhimen Hospital, Beijing
Other Study IDs: 2022YFC3501104-01
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke, Acute
Keywords: Shuxuetong Injection; Intravenous Thrombolysis; Patient Registry
MeSH Terms: conditions — Ischemic Stroke | interventions — shuxuetong

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: The exposure group was defined as patients receiving Shuxuetong injection and guideline-standardized treatment after intravenous alteplase or tenecteplase.
  Mainly based on the following guidelines:(1)Guidelines for the diagnosis and treatment of acute ischemic stroke in China 2018; (2)Guidelines for secondary prevention of ischemic stroke and transient ischemic attack in China 2022.
  Interventions: Drug: Shuxuetong Injection
- Non-exposure group: The non-exposed group was defined as patients receiving guideline-standardized treatment after intravenous alteplase or tenecteplase.

INTERVENTIONS:
Drug: Shuxuetong Injection — According to clinical real treatment records
  Groups: Exposure group

SUMMARY:
Acute ischemic stroke is one of the main diseases leading to high risk of disability and morbidity worldwide. Since intravenous thrombolysis(IVT) can effectively improve the long-term functional prognosis of acute ischemic stroke(AIS), IVT within 4.5 hours of onset has been widely recommended by international guidelines.

Although 35-53% of AIS patients achieve functional independence after receiving IVT, there are still a large number of patients who are disabled or even dead, and nearly 70% of patients have ineffective recanalization. Therefore, there is an urgent need for therapeutic drugs after IVT to further improve the prognosis and reduce the burden of AIS.

Shuxuetong injection is widely used in China in patients with AIS after IVT, but the situation in real clinical practice is unclear. Therefore, the study aims to evaluate the effectiveness and safety of Shuxuetong Injection in patients with AIS treated with intravenous alteplase and tenecteplase, and obtain high-quality clinical evidence.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged ≥18 years
* Diagnosis of acute ischemic stroke
* Receiving alteplase or tenecteplase treatment ≤ 4.5 hours of onset
* Signed informed consent by patient or legally authorized representatives

Exclusion Criteria:

* Having received or planing to undergo endovascular therapy (including mechanical thrombectomy, arterial thrombolysis, angioplasty, etc.)
* Life expectancy is less than 90 days
* Other factors that the researchers think are not suitable for participating in the research
* Currently receiving any experimental treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke who received alteplase or tenecteplase within 4.5 hours of onset
Sampling Method: Non-Probability Sample
Enrollment: 2008 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of mRS (0-1) | 90±7 days
  The modified Rankin Scale (mRS) score ranges from 0 (best score) to 6 (worst score).

SECONDARY OUTCOMES:
Proportion of mRS (0-2) | 90±7 days
Proportion of mRS (0-1) or returning to baseline | 90±7 days
Distribution of mRS | 90±7 days
Change of NIHSS | baseline, 14 days or the day of discharge
  The change in the National Institute of Health Stroke Scale (NIHSS) scores from baseline to 14 days or the day of discharge. The NIHSS score ranges from 0 (best score) to 42 (worst score).
BI | 90±7 days
  The Barthel Index (BI) score ranges from 0 (worst score) to 100 (best score).
Total mortality | Within 90 days
  The occurrence of mortality of any cause within 90 days.
Serious Adverse Events | Within 90 days
  The occurrence of serious adverse events including any event resulting in prolonged hospital time, permanent damage to the body system or organ, a life-threatening condition or death within 90 days.

CONTACTS AND LOCATIONS:
Locations (78):
- China (78):
  - Beijing Royal Integrative Medicine Hospital, Beijing, Beijing Municipality
  - China Aerospace Science and Industry Corporation 731 Hospital, Beijing, Beijing Municipality
  - Chongqing Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - University-Town Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Nanning First People's Hospital, Nanning, Guangxi
  - Guizhou People's Hospital, Guiyang, Guizhou
  - Hebei CangZhou Hospital of Integrated Traditional Chinese and Western Medicine, Cangzhou, Hebei
  - Tangshan Central Hospital, Tangshan, Hebei
  - The First Affiliated Hospital Of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hongqi Hospital Affiliated to Mudanjiang Medical University, Mudanjiang, Heilongjiang
  - Anyang Third People's Hospital, Anyang, Henan
  - Huaxian People's Hospital, Anyang, Henan
  - Neihuang People's Hospital, Anyang, Henan
  - Jiaozuo Second People's Hospital, Jiaozuo, Henan
  - Kaifeng People's Hospital, Kaifeng, Henan
  - Luohe Sixth People's Hospital, Luohe, Henan
  - Nanyang Nanshi Hospital, Nanyang, Henan
  - Baofeng Chinese Medicine Hospital, Pingdingshan, Henan
  - Baofeng People's Hospital, Pingdingshan, Henan
  - Pingdingshan First People's Hospital, Pingdingshan, Henan
  - Ye County People's Hospital, Pingdingshan, Henan
  - Shangqiu Municipal Hospital, Shangqiu, Henan
  - Changyuan Chinese Medicine Hospital, Xinxiang, Henan
  - The First Affiliated Hospital Of Xinxiang Medical University, Xinxiang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Xinxiang First People's Hospital, Xinxiang, Henan
  - Xi County Central Hospital, Xinyang, Henan
  - The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan
  - Runan People's Hospital, Zhumadian, Henan
  - Changsha First Hospital, Changsha, Hunan
  - The Affiliated Hospital of Hunan Academy of Chinese Medicine, Changsha, Hunan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Hunan
  - Nanjing Chinese Medicine Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Pengzhou Chinese Medicine Hospital, Pengzhou, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - Gaoxin Hospital Of The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Jiangxi People's Hospital, Nanchang, Jiangxi
  - Jilin Central General Hospital, Jilin, Jilin
  - Songyuan Jilin Oifield Hospital, Songyuan, Jilin
  - Anshan Central Hospital, Anshan, Liaoning
  - 967 Hospital of The Joint Logistics Support Force of PLA, Dalian, Liaoning
  - Central Hospital Affiliated Dalian University of Technology, Dalian, Liaoning
  - Dalian University Affiliated Xinhua Hospital, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Jinzhou Central Hospital, Jinzhou, Liaoning
  - Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Tieling Central Hospital, Tieling, Liaoning
  - Binzhou Medical University Hospital/ The First School of Clinical Medicine of Binzhou Medical University, Binzhou, Shandong
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Liaocheng Third People's Hospital, Liaocheng, Shandong
  - Linyi Hospital of Traditional Chinese Medicine, Linyi, Shandong
  - Ningjin People's Hospital, Ningjin, Shandong
  - Qingdao Huangdao District Chinese Medicine Hospital, Qingdao, Shandong
  - Weihai Wendeng District People's Hospital, Weihai, Shandong
  - Zibo First Hospital, Zibo, Shandong
  - Zibo Hospital of Traditional Chinese Medicine, Zibo, Shandong
  - Shanghai Pingdingshan Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Affiliated Hospital Of Changzhi Institute Of TCM, Changzhi, Shanxi
  - Gujiao Central Hospital, Taiyuan, Shanxi
  - Chengdu Integrated TCM & Western Medicine Hospital, Chengdu, Sichuan
  - Chengdu Seventh People's Hospital, Chengdu, Sichuan
  - Chengdu Shuangliu District Chinese Medicine Hospital, Chengdu, Sichuan
  - Chengdu Xinjin District Chinese Medicine Hospital, Chengdu, Sichuan
  - Jintang Second People's Hospital, Chengdu, Sichuan
  - Sichuan Tianfu People's Hospital, Chengdu, Sichuan
  - The Fourth People's Hospital of Sichuan Province, Chengdu, Sichuan
  - Xuyong Chinese Medicine Hospital, Luzhou, Sichuan
  - Qingshen People's Hospital, Meishan, Sichuan
  - Mianyang Third People's Hospital, Mianyang, Sichuan
  - Nanchong Central Hospital, Nanchong, Sichuan
  - Panzhihua Central Hospital, Panzhihua, Sichuan
  - Yibin Chinese Medicine Hospital, Yibin, Sichuan
  - Beijing University of Chinese Medicine Affiliated Dongzhimen Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided